CLINICAL TRIAL: NCT02817841
Title: A Multicenter, Open-label, Single-Arm Study to Evaluate the Contraceptive Efficacy and Safety of a Combined Oral Contraceptive Containing 15 mg Estetrol and 3 mg Drospirenone
Brief Title: E4 FREEDOM (Female Response Concerning Efficacy and Safety of Estetrol/Drospirenone as Oral Contraceptive in a Multicentric Study) - United States/Canada Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estetra (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MIT-Es0001-C302
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-10

CONDITIONS: Contraception
Keywords: Estetrol; Drospirenone; Prevention of pregnancy; Oral contraception
MeSH Terms: interventions — Estetrol; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 15 mg E4/3 mg DRSP (Experimental): 15 mg estetrol (E4)/3 mg drospirenone (DRSP) combined oral contraceptive
  Interventions: Drug: 15 mg E4/3 mg DRSP

INTERVENTIONS:
Drug: 15 mg E4/3 mg DRSP — 15 mg estetrol and 3 mg drospirenone tablets administered once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
  Other Names: 15 mg estetrol and 3 mg drospirenone

SUMMARY:
The objectives of this study are to evaluate the contraceptive efficacy, vaginal bleeding pattern (cycle control), and the general safety and acceptability of the 15 mg estetrol (E4)/3 mg drospirenone (DRSP) combination in healthy women aged 16 to 50 years.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexually active female at risk for pregnancy and requesting contraception.
* Negative serum pregnancy test at subject screening.
* Willing to use the investigational product as the primary method of contraception for 13 consecutive cycles.
* Good physical and mental health on the basis of medical, surgical and gynecological history, physical examination, gynecological examination, clinical laboratory, and vital signs.
* Body mass index (BMI) below or equal to (≤) 35.0 kg/m2.
* Able to fulfill the requirements of the protocol and have indicated a willingness to participate in the study by providing written informed consent.
* Willing and able to complete the diaries and questionnaires.

Exclusion Criteria:

* Known hypersensitivity to any of the investigational product ingredients.
* Smoking if ≥ 35 years old, at screening.
* Any condition associated with decrease fertility.
* Dyslipoproteinemia requiring active treatment with antilipidemic agent.
* Diabetes mellitus with vascular involvement (nephropathy, retinopathy, neuropathy, other) or diabetes mellitus of more than 20-year duration.
* Arterial hypertension.
* Any condition associated with an increased risk of venous thromboembolism and/or arterial thromboembolism.
* Any condition associated with abnormal uterine/vaginal bleeding.
* Abnormal Pap test based on current international recommendations.
* Presence of an undiagnosed breast mass.
* Current symptomatic gallbladder disease.
* History of combined oral contraceptive (COC) related cholestasis.
* Presence or history of severe hepatic disease.
* Presence or history of pancreatitis if associated with hypertriglyceridemia.
* Porphyria.
* Presence or history of hepatocellular adenoma or malignant liver tumors.
* Renal impairment.
* Hyperkaliemia or presence of conditions that predispose to hyperkaliemia.
* Presence or history of hormone-related malignancy.
* History of non-hormone-related malignancy within 5 years before screening. Subjects with a non-melanoma skin cancer are allowed in the study.
* History of alcohol or drug abuse (including laxatives) within 12 months prior to screening.
* Use of drugs potentially triggering interactions with COCs.
* Any condition that could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the investigational product.
* Uncontrolled thyroid disorders.
* Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last 3 months (90 days) prior to study entry. Subjects who participated in an oral contraceptive clinical study, using FDA/European (EU) approved active ingredients, may be enrolled 2 months (60 days) after completing the preceding study.
* Sponsor, Contract Research Organization (CRO) or Investigator's site personnel directly affiliated with this study.
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2148 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estetra, Study Director — Estetra
Locations (2):
- Thomas Jefferson University Obstetrics and Gynecology, Philadelphia, Pennsylvania, United States
- Clinique de Santé des Femmes, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creinin MD, Jensen JT, Chen MJ, Black A, Costescu D, Foidart JM. Combined Oral Contraceptive Adherence and Pregnancy Rates. Obstet Gynecol. 2023 May 1;141(5):989-994. doi: 10.1097/AOG.0000000000005155. Epub 2023 Apr 5. PMID 37023457

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2,148 participants aged 16-50 years were enrolled. Of those, 1,864 participants started the investigational product. Two hundred and eighty-four participants did not start the investigational product for the following reasons: lost to follow-up (166), withdrew consent (31), and other reasons (87).
Period: Overall Study
Arm/Group | 15 mg E4/3 mg DRSP
Started | 1864
Completed | 1016
Not Completed | 848
Not completed — Lost to Follow-up | 287
Not completed — Withdrawal by Subject | 183
Not completed — Adverse event not related to bleeding | 131
Not completed — Adverse event related to bleeding | 51
Not completed — Pregnancy | 32
Not completed — Pregnancy wish | 17
Not completed — Other reasons | 53
Not completed — Protocol Violation | 94

BASELINE CHARACTERISTICS:
Population: All participants aged 16 to 50 years who received at least one dose of 15 mg E4/3 mg DRSP
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74
  Between 18 and 65 years | 1,790
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (6.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1,864
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 488
  Not Hispanic or Latino | 1,376
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 152
  United States | 1,712
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 25.89 (4.705)

OUTCOME MEASURES:

1. Primary Outcome: The Number of On-treatment Pregnancies (With + 7-day Window) Per 100 Woman-years of Exposure (Pearl Index) in Subjects Aged 16 to 35 Years, Inclusive, at the Time of Screening
Description: On-treatment pregnancies are pregnancies with an estimated date of conception within the in-treatment period i.e. Day 1 to 7 days after the last intake of investigational product (whether active or inactive tablet). The Pearl Index, defined as the number of pregnancies per 100 women-years of treatment was calculated as: Pearl Index = (1300*number of on-treatment pregnancies)/number of women 28-day equivalent cycles of treatment. Only at-risk cycles were included in the denominator of the Pearl Index calculation, unless a conception occurred during a cycle.
  At-risk-cycle was defined as cycle in which no other methods of birth control (including condoms and emergency contraception) were used by the subject as confirmed in the subject diary and during which the subject confirmed that sexual intercourse had occurred.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 35 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,524
Pearl Index | 2.65 [1.73 to 3.88]

2. Secondary Outcome: The Number of On-treatment Pregnancies (With +7-day Window) as Assessed by the Method Failure Pearl Index in Subjects Aged 16 to 35 Years, Inclusive, at the Time of Screening
Description: On-treatment pregnancies are pregnancies with an estimated date of conception within the in-treatment period i.e. Day 1 to 7 days after the last intake of investigational product (whether active or inactive tablet). The method failure Pearl Index, defined as the number of pregnancies as a result of method failure per 100 women-years of treatment, was calculated as follow: (1300*number of on-treatment pregnancies as a result of method failure)/number of women 28-day equivalent cycles of treatment. Pregnancies due to user failure were excluded from the numerator. User failure pregnancies were pregnancies that occurred when the subject did not take the investigational product correctly.
  At-risk-cycle was defined as cycle in which no other methods of birth control (including condoms and emergency contraception) were used by the subject and during which the subject confirmed that sexual intercourse had occurred.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 35 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Method failure Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,524
Method failure Pearl Index | 1.43 [0.78 to 2.39]

3. Secondary Outcome: The Number of On-treatment Pregnancies (With + 7-day Window) Per 100 Woman-years of Exposure (Pearl Index) in the Overall Study Population (16-50 Years)
Description: as for outcome 1
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,705
Pearl Index | 2.52 [1.68 to 3.64]

4. Secondary Outcome: The Number of On-treatment Pregnancies as Assessed by the Method Failure Pearl Index in the Overall Study Population (16-50 Years)
Description: as for outcome 2
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Method failure Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,705
Method failure Pearl Index | 1.44 [0.82 to 2.34]

5. Secondary Outcome: Rate of Pregnancy (Life-table Analysis) in Participants Aged 16 to 35 Years
Description: The life-table analysis evaluates the cumulative probability of pregnancy over 13 cycles. Cumulative Rate and 95% CI are from Kaplan-Meier estimation. Only on-treatment pregnancies are included.
  On-treatment pregnancy is a pregnancy with an estimated date of conception after the date of the first dose of study medication to 7 days after the last dose of study medication (regardless of whether the last dose is an active or inactive tablet) inclusive.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 35 years, inclusive, at screening, who received at least one dose of investigational product
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 901
percentage of participants | 2.06 [1.40 to 3.04]

6. Secondary Outcome: Rate of Pregnancy (Life-table Analysis) in Participants Aged 16 to 50 Years
Description: The life-table analysis evaluates the cumulative probability of pregnancy over 13 cycles. Cumulative Rate and 95% confidence interval (CI) are from Kaplan-Meier estimation. Only on-treatment pregnancies are included.
  On-treatment pregnancy is a pregnancy with an estimated date of conception after the date of the first dose of study medication to 7 days after the last dose of study medication (regardless of whether the last dose is an active or inactive tablet) inclusive.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, who received at least one dose of investigational product
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,017
percentage of participants | 2.00 [1.38 to 2.91]

7. Secondary Outcome: Number of Subjects With Unscheduled Bleeding/Spotting Episodes
Description: Unscheduled bleeding/spotting is defined as any bleeding/spotting that occurs while taking active hormones that does not meet the criteria for scheduled bleeding.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants
  Cycle 1: number analyzed (Participants) | 1,758
  Cycle 1 | 532
  Cycle 2: number analyzed (Participants) | 1,579
  Cycle 2 | 345
  Cycle 3: number analyzed (Participants) | 1,526
  Cycle 3 | 337
  Cycle 4: number analyzed (Participants) | 1,420
  Cycle 4 | 302
  Cycle 5: number analyzed (Participants) | 1,352
  Cycle 5 | 238
  Cycle 6: number analyzed (Participants) | 1,319
  Cycle 6 | 253
  Cycle 7: number analyzed (Participants) | 1,235
  Cycle 7 | 229
  Cycle 8: number analyzed (Participants) | 1,208
  Cycle 8 | 204
  Cycle 9: number analyzed (Participants) | 1,162
  Cycle 9 | 221
  Cycle 10: number analyzed (Participants) | 1,053
  Cycle 10 | 184
  Cycle 11: number analyzed (Participants) | 1,028
  Cycle 11 | 159
  Cycle 12: number analyzed (Participants) | 1,006
  Cycle 12 | 175

8. Secondary Outcome: Number of Unscheduled Bleeding Days Per Cycle
Description: Unscheduled bleeding is defined as any bleeding that occurs while taking active hormones that does not meet the criteria for scheduled bleeding and/or spotting.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Days
  Cycle 1: number analyzed (Participants) | 1,758
  Cycle 1 | 0.4 (1.42)
  Cycle 2: number analyzed (Participants) | 1,579
  Cycle 2 | 0.3 (1.08)
  Cycle 3: number analyzed (Participants) | 1,526
  Cycle 3 | 0.4 (1.20)
  Cycle 4: number analyzed (Participants) | 1,420
  Cycle 4 | 0.3 (1.00)
  Cycle 5: number analyzed (Participants) | 1,352
  Cycle 5 | 0.3 (1.04)
  Cycle 6: number analyzed (Participants) | 1,319
  Cycle 6 | 0.3 (1.04)
  Cycle 7: number analyzed (Participants) | 1,235
  Cycle 7 | 0.3 (1.04)
  Cycle 8: number analyzed (Participants) | 1,208
  Cycle 8 | 0.2 (0.94)
  Cycle 9: number analyzed (Participants) | 1,162
  Cycle 9 | 0.3 (1.01)
  Cycle 10: number analyzed (Participants) | 1,053
  Cycle 10 | 0.3 (1.07)
  Cycle 11: number analyzed (Participants) | 1,028
  Cycle 11 | 0.2 (0.94)
  Cycle 12: number analyzed (Participants) | 1,006
  Cycle 12 | 0.2 (0.98)

9. Secondary Outcome: Number of Unscheduled Spotting Days Per Cycle
Description: Unscheduled spotting is defined as any spotting that occurs while taking active hormones that does not meet the criteria for scheduled bleeding and/or spotting.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Days
  Cycle 1: number analyzed (Participants) | 1,758
  Cycle 1 | 1.0 (2.21)
  Cycle 2: number analyzed (Participants) | 1,579
  Cycle 2 | 0.6 (1.50)
  Cycle 3: number analyzed (Participants) | 1,526
  Cycle 3 | 0.6 (1.40)
  Cycle 4: number analyzed (Participants) | 1,420
  Cycle 4 | 0.5 (1.31)
  Cycle 5: number analyzed (Participants) | 1,352
  Cycle 5 | 0.5 (1.26)
  Cycle 6: number analyzed (Participants) | 1,319
  Cycle 6 | 0.5 (1.30)
  Cycle 7: number analyzed (Participants) | 1,235
  Cycle 7 | 0.5 (1.31)
  Cycle 8: number analyzed (Participants) | 1,208
  Cycle 8 | 0.4 (1.18)
  Cycle 9: number analyzed (Participants) | 1,162
  Cycle 9 | 0.5 (1.21)
  Cycle 10: number analyzed (Participants) | 1,053
  Cycle 10 | 0.4 (1.20)
  Cycle 11: number analyzed (Participants) | 1,028
  Cycle 11 | 0.4 (1.08)
  Cycle 12: number analyzed (Participants) | 1,006
  Cycle 12 | 0.4 (1.09)

10. Secondary Outcome: Number of Subjects With Absence of Scheduled Bleeding and/or Spotting
Description: Scheduled bleeding/spotting is defined as any bleeding/spotting that occurs during the hormone-free interval (i.e. Days 25 - 28) and continues through Days 1-3 of the subsequent active cycle.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants
  Cycle 1: number analyzed (Participants) | 1,758
  Cycle 1 | 230
  Cycle 2: number analyzed (Participants) | 1,579
  Cycle 2 | 254
  Cycle 3: number analyzed (Participants) | 1,526
  Cycle 3 | 274
  Cycle 4: number analyzed (Participants) | 1,420
  Cycle 4 | 233
  Cycle 5: number analyzed (Participants) | 1,352
  Cycle 5 | 209
  Cycle 6: number analyzed (Participants) | 1,319
  Cycle 6 | 225
  Cycle 7: number analyzed (Participants) | 1,235
  Cycle 7 | 191
  Cycle 8: number analyzed (Participants) | 1,208
  Cycle 8 | 183
  Cycle 9: number analyzed (Participants) | 1,162
  Cycle 9 | 180
  Cycle 10: number analyzed (Participants) | 1,053
  Cycle 10 | 137
  Cycle 11: number analyzed (Participants) | 1,028
  Cycle 11 | 136
  Cycle 12: number analyzed (Participants) | 1,006
  Cycle 12 | 134

11. Secondary Outcome: Number of Scheduled Bleeding and/or Spotting Days Per Cycle
Description: as for outcome 10
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Days
  Cycle 1: number analyzed (Participants) | 1,758
  Cycle 1 | 6.1 (10.16)
  Cycle 2: number analyzed (Participants) | 1,579
  Cycle 2 | 4.7 (4.01)
  Cycle 3: number analyzed (Participants) | 1,526
  Cycle 3 | 4.7 (6.72)
  Cycle 4: number analyzed (Participants) | 1,420
  Cycle 4 | 4.8 (6.50)
  Cycle 5: number analyzed (Participants) | 1,352
  Cycle 5 | 4.4 (3.70)
  Cycle 6: number analyzed (Participants) | 1,319
  Cycle 6 | 4.4 (3.39)
  Cycle 7: number analyzed (Participants) | 1,235
  Cycle 7 | 4.5 (5.00)
  Cycle 8: number analyzed (Participants) | 1,208
  Cycle 8 | 4.5 (3.69)
  Cycle 9: number analyzed (Participants) | 1,162
  Cycle 9 | 4.4 (5.64)
  Cycle 10: number analyzed (Participants) | 1,053
  Cycle 10 | 4.3 (3.41)
  Cycle 11: number analyzed (Participants) | 1,028
  Cycle 11 | 4.3 (3.87)
  Cycle 12: number analyzed (Participants) | 1,006
  Cycle 12 | 4.3 (3.07)

12. Secondary Outcome: Number of Subjects With Bleeding and/or Spotting Episodes by Reference Period
Description: Bleeding data were analysed by 91-day reference period. There were 4 RPs: Reference Period 1 = Day 1 to Day 91; Reference Period 2 = Day 92 to Day 182; Reference Period 3 = Day 183 to Day 273; and Reference Period 4 = Day 274 to Day 364.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable reference period for the bleeding analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 15 mg E4/3 mg DRSP - RP1: 15 mg estetrol (E4)/3 mg drospirenone (DRSP) combined oral contraceptive
  15 mg E4/3 mg DRSP: 15 mg estetrol and 3 mg drospirenone tablets administered once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
Arm/Group | 15 mg E4/3 mg DRSP - RP1
Number analyzed (Participants) | 1,864
Participants
  Reference Period 1 | 1,249
  Reference Period 2: number analyzed (Participants) | 1,120
  Reference Period 2 | 1,098
  Reference Period 3: number analyzed (Participants) | 1,002
  Reference Period 3 | 982
  Reference Period 4: number analyzed (Participants) | 933
  Reference Period 4 | 914

13. Secondary Outcome: Mean Number of Bleeding and Spotting Days by Reference Period
Description: Bleeding data were analysed by 91-day reference period (RP). There were 4 RPs: Reference Period 1 = Day 1 to Day 91; Reference Period 2 = Day 92 to Day 182; Reference Period 3 = Day 183 to Day 273; and Reference Period 4 = Day 274 to Day 364.
Time Frame: up to 12 months (13 cycles)
Population: Participants aged 16 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Days
  Reference Period 1 | 3.6 (1.23)
  Reference Period 2: number analyzed (Participants) | 1,120
  Reference Period 2 | 3.3 (1.27)
  Reference Period 3: number analyzed (Participants) | 1,002
  Reference Period 3 | 3.3 (1.25)
  Reference Period 4: number analyzed (Participants) | 933
  Reference Period 4 | 3.9 (1.30)

14. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability.
Description: A treatment-emergent adverse event (TEAE) was defined as any AE not present prior to the initiation of the treatment or any event already present that worsened in either intensity or frequency following exposure to the treatment. Since the starting point for adverse event (AE) collection was the signing of the informed consent, not the start of the investigational product, the AEs recorded prior to first investigational product administration were designated as AEs while those that occurred or worsened after the initiation of the investigational product were designated as TEAEs.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants | 1,002

15. Secondary Outcome: Number of Participants With Clinically Significant out-of Range Hematology Results
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants | 8

16. Secondary Outcome: Number of Participants With Clinically Significant out-of Range Serum Chemistry and Lipid Profile Results
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants | 21

17. Secondary Outcome: Number of Subjects With Clinically Abnormal Vital Signs
Description: Vital signs included sitting systolic and diastolic blood pressures, and heart rate. All abnormal findings in vital signs that were considered by the Investigator to be clinically significant were recorded as adverse events.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants | 10

18. Secondary Outcome: Number of Participants With Clinically Abnormal Physical Examination Results
Description: Physical examinations included an evaluation of body as a whole, skin, head, eyes, ears, nose, and throat, neck, cardiovascular, respiratory, musculoskeletal, neurologic, lymphatic/thyroid, abdomen. When reporting the results of the physical examination, the use of the "Abnormal" category was reserved for findings that were considered clinically significant, in the opinion of the Investigator; the "Normal" category included "Abnormal" results that were not clinically significant, as well as no findings.
Time Frame: Baseline and end of treatment (Cycle 13 with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening, who received at least one dose of investigational product with baseline and end of treatment (EOT) data.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants
  Body as a whole -Baseline: Normal | 1,862
  Body as a whole -Baseline: Abnormal | 2
  Body as a whole -Baseline: Not done | 0
  Body as a whole - EOT: number analyzed (Participants) | 1,432
  Body as a whole - EOT: Normal | 1,431
  Body as a whole - EOT: Abnormal | 0
  Body as a whole - EOT: Not done | 1
  Skin - Baseline: Normal | 1,838
  Skin - Baseline: Abnormal | 25
  Skin - Baseline: Not done | 1
  Skin - EOT: number analyzed (Participants) | 1,431
  Skin - EOT: Normal | 1,412
  Skin - EOT: Abnormal | 18
  Skin - EOT: Not done | 1
  Head, Eyes, Ears, Nose and Throat - Baseline: Normal | 1,856
  Head, Eyes, Ears, Nose and Throat - Baseline: Abnormal | 7
  Head, Eyes, Ears, Nose and Throat - Baseline: Not done | 1
  Head, Eyes, Ears, Nose - EOT: number analyzed (Participants) | 1,432
  Head, Eyes, Ears, Nose - EOT: Normal | 1,424
  Head, Eyes, Ears, Nose - EOT: Abnormal | 2
  Head, Eyes, Ears, Nose - EOT: Not done | 6
  Neck - Baseline: Normal | 1,852
  Neck - Baseline: Abnormal | 2
  Neck - Baseline: Not done | 10
  Neck - EOT: number analyzed (Participants) | 1,432
  Neck - EOT: Normal | 1,429
  Neck - EOT: Abnormal | 3
  Neck - EOT: Not done | 0
  Cardiovascular - Baseline: Normal | 1,862
  Cardiovascular - Baseline: Abnormal | 2
  Cardiovascular - Baseline: Not done | 0
  Cardiovascular - EOT: number analyzed (Participants) | 1,432
  Cardiovascular - EOT: Normal | 1,429
  Cardiovascular - EOT: Abnormal | 3
  Cardiovascular - EOT: Not done | 0
  Respiratory - Baseline: Normal | 1,861
  Respiratory - Baseline: Abnormal | 3
  Respiratory - Baseline: Not done | 0
  Respiratory - EOT: number analyzed (Participants) | 1,432
  Respiratory - EOT: Normal | 1,428
  Respiratory - EOT: Abnormal | 1
  Respiratory - EOT: Not done | 3
  Musculoskeletal - Baseline: Normal | 1,852
  Musculoskeletal - Baseline: Abnormal | 2
  Musculoskeletal - Baseline: Not done | 10
  Musculoskeletal - EOT: number analyzed (Participants) | 1,432
  Musculoskeletal - EOT: Normal | 1,423
  Musculoskeletal - EOT: Abnormal | 3
  Musculoskeletal - EOT: Not done | 6
  Neurologic - Baseline: Normal | 1,851
  Neurologic - Baseline: Abnormal | 1
  Neurologic - Baseline: Not done | 12
  Neurologic - EOT: number analyzed (Participants) | 1,432
  Neurologic - EOT: Normal | 1,423
  Neurologic - EOT: Abnormal | 1
  Neurologic - EOT: Not done | 8
  Lymphatic/Thyroid - Baseline: Normal | 1,860
  Lymphatic/Thyroid - Baseline: Abnormal | 4
  Lymphatic/Thyroid - Baseline: Not done | 0
  Lymphatic/Thyroid - EOT: number analyzed (Participants) | 1,432
  Lymphatic/Thyroid - EOT: Normal | 1,431
  Lymphatic/Thyroid - EOT: Abnormal | 1
  Lymphatic/Thyroid - EOT: Not done | 0
  Abdomen - Baseline: Normal | 1,860
  Abdomen - Baseline: Abnormal | 3
  Abdomen - Baseline: Not done | 1
  Abdomen - EOT: number analyzed (Participants) | 1,432
  Abdomen - EOT: Normal | 1,431
  Abdomen - EOT: Abnormal | 1
  Abdomen - EOT: Not done | 0
  Additional findings -Baseline: number analyzed (Participants) | 25
  Additional findings -Baseline: Normal | 3
  Additional findings -Baseline: Abnormal | 1
  Additional findings -Baseline: Not done | 21
  Additional findings - EOT: number analyzed (Participants) | 34
  Additional findings - EOT: Normal | 3
  Additional findings - EOT: Abnormal | 1
  Additional findings - EOT: Not done | 30

19. Secondary Outcome: Number of Participants With Clinically Abnormal Gynecological Examination Results
Description: Gynecological examinations included breast examination (performed by palpation) and assessment of the adnexa, cervix, uterus, vagina, and external genitalia.
  When reporting the results, the use of the "Abnormal" category was reserved for findings that were considered clinically significant, in the opinion of the Investigator; the "Normal" category included "Abnormal" results that were not clinically significant, as well as no findings.
Time Frame: Baseline and end of treatment (Cycle 13 with 1 cycle = 28 days)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Participants
  Breast -Baseline: Normal | 1,857
  Breast -Baseline: Abnormal | 6
  Breast -Baseline: Not done | 1
  Breast - EOT: number analyzed (Participants) | 1,414
  Breast - EOT: Normal | 1,387
  Breast - EOT: Abnormal | 16
  Breast - EOT: Not done | 11
  Adnexa - Baseline: Normal | 1,861
  Adnexa - Baseline: Abnormal | 1
  Adnexa - Baseline: Not done | 2
  Adnexa - EOT: number analyzed (Participants) | 1,414
  Adnexa - EOT: Normal | 1,404
  Adnexa - EOT: Abnormal | 4
  Adnexa - EOT: Not done | 6
  Cervix- Baseline: Normal | 1,862
  Cervix- Baseline: Abnormal | 2
  Cervix- Baseline: Not done | 0
  Cervix - EOT: number analyzed (Participants) | 1,414
  Cervix - EOT: Normal | 1,397
  Cervix - EOT: Abnormal | 5
  Cervix - EOT: Not done | 12
  Uterus - Baseline: Normal | 1,861
  Uterus - Baseline: Abnormal | 3
  Uterus - Baseline: Not done | 0
  Uterus - EOT: number analyzed (Participants) | 1,414
  Uterus - EOT: Normal | 1,402
  Uterus - EOT: Abnormal | 7
  Uterus - EOT: Not done | 5
  Vagina - Baseline: Normal | 1,841
  Vagina - Baseline: Abnormal | 23
  Vagina - Baseline: Not done | 0
  Vagina - EOT: number analyzed (Participants) | 1,414
  Vagina - EOT: Normal | 1,386
  Vagina - EOT: Abnormal | 22
  Vagina - EOT: Not done | 6
  External genitalia - Baseline: Normal | 1,860
  External genitalia - Baseline: Abnormal | 4
  External genitalia - Baseline: Not done | 0
  External genitalia - EOT: number analyzed (Participants) | 1,413
  External genitalia - EOT: Normal | 1,398
  External genitalia - EOT: Abnormal | 10
  External genitalia - EOT: Not done | 5

20. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Results at Baseline and End of Treatment - Percentage Maximum (Sum of First 14 Items)
Description: The Q-LES-Q-SF is a self-report measure designed to assess the degree of enjoyment and satisfaction in daily functioning. Participants were asked to rate 16 different items on a 5-point scale where score 1 = very poor and score 5 = very good. A raw total score is calculated by summing the first 14 items and ranges from 14 to 70. The raw total score is then transformed into a percentage maximum score using the following formula: (raw total score-minimum score)/(maximum possible raw score-minimum score). The minimum raw is 14 and maximum raw score is 70. Thus the formula for % maximum score can be written as (raw score -14)/56. A higher percentage maximum score indicates a higher life enjoyment and satisfaction.
Time Frame: Baseline and end of treatment (Cycle 13 with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening with baseline and end of treatment (EOT) Q-LES-Q-SF results.
Measure: Mean (Standard Deviation); unit: Percentage maximum score on a scale
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Percentage maximum score on a scale
  Baseline: number analyzed (Participants) | 1,490
  Baseline | 75.8 (13.58)
  EOT: number analyzed (Participants) | 1,358
  EOT | 75.4 (14.80)

21. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Results at Baseline and End of Treatment - Satisfaction With Medicine and Overall Life Satisfaction and Contentment Over the Past Week
Description: The Q-LES-Q-SF is a self-report measure designed to assess the degree of enjoyment and satisfaction in daily functioning. Participants were asked to rate 16 different items on a 5-point scale where score 1 = very poor and score 5 = very good. The last two items - item 15 rating "satisfaction with medicine" and item 16 rating "overall life satisfaction over the past week" are two global items that are scored individually. For both items, a higher score is associated with a better outcome.
Time Frame: Baseline and end of treatment (Cycle 13 with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening with baseline and end of treatment (EOT) Q-LES-Q-SF results.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,864
Units on a scale
  Satisfaction with medicine - Baseline: number analyzed (Participants) | 493
  Satisfaction with medicine - Baseline | 4.2 (0.69)
  Satisfaction with medicine - EOT: number analyzed (Participants) | 514
  Satisfaction with medicine - EOT | 4.1 (0.75)
  Overall life satisfaction - Baseline: number analyzed (Participants) | 1,490
  Overall life satisfaction - Baseline | 4.1 (0.73)
  Overall life satisfaction - EOT: number analyzed (Participants) | 1,358
  Overall life satisfaction - EOT | 4.1 (0.77)

22. Secondary Outcome: Change From Baseline to End of Treatment in the Score of the Menstrual Distress Questionnaire (MDQ)
Description: The MDQ is a standard method for measuring cyclical perimenstrual symptoms. The participants rated common symptoms and feelings associated with menstruation using the following scale: 0 (no experience of symptom), 1 (present, mild), 2 (present, moderate), 3 (present, strong),and 4 (present, severe) observed during pre-menstrual (4 days before menstruation), menstrual (most recent flow) and intermenstrual (remainder of the cycle) phases. Reported values are values at Cycle 13 minus values at Baseline. An overall positive change from baseline represents an increase in symptom or feeling severity.
Time Frame: Baseline and end of treatment (Cycle 13 with 1 cycle = 28 days)
Population: Participants aged 16 to 50 years, inclusive, at screening with both baseline and end of treatment (EOT) MDQ results
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 15 mg E4/3 mg DRSP - Intermenstrual Phase; 15 mg E4/3 mg DRSP - Premenstrual Phase; 15 mg E4/3 mg DRSP - Menstrual Phase: 15 mg estetrol (E4)/3 mg drospirenone (DRSP) combined oral contraceptive
  15 mg E4/3 mg DRSP: 15 mg estetrol and 3 mg drospirenone tablets administered once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
Arm/Group | 15 mg E4/3 mg DRSP - Intermenstrual Phase | 15 mg E4/3 mg DRSP - Premenstrual Phase | 15 mg E4/3 mg DRSP - Menstrual Phase
Number analyzed (Participants) | 1,864 | 1,864 | 1,864
units on a scale
  Pain: number analyzed (Participants) | 1,304 | 1,297 | 1,302
  Pain | -0.3 (4.13) | -0.1 (4.19) | -0.6 (4.68)
  Water retention: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Water retention | -0.1 (2.58) | -0.2 (2.91) | -0.2 (2.9)
  Autonomic reactions: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Autonomic reactions | 0.0 (1.56) | 0.0 (1.69) | 0.1 (1.71)
  Negative affect: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Negative affect | -0.1 (5.17) | -0.4 (5.94) | -0.3 (5.98)
  Impaired concentration: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Impaired concentration | 0.0 (3.00) | -0.1 (3.19) | -0.1 (3.42)
  Behaviour change: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Behaviour change | -0.0 (2.99) | -0.0 (3.19) | -0.0 (3.37)
  Arousal: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Arousal | -0.2 (4.66) | -0.2 (4.42) | -0.2 (4.28)
  Control: number analyzed (Participants) | 1,305 | 1,298 | 1,303
  Control | 0.1 (1.69) | 0.1 (1.94) | 0.1 (1.92)

ADVERSE EVENTS:
Time Frame: From screening to end of treatment (13 months)
Arm/Group | 15 mg E4/3 mg DRSP
All-Cause Mortality (participants affected / at risk) | 1/1864
Serious Adverse Events (participants affected / at risk) | 25/1864
Other Adverse Events (participants affected / at risk) | 1002/1864
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg E4/3 mg DRSP (N=1864)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 7 (7)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Affective disorder (Psychiatric disorders) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1)
Infection parasitic (Infections and infestations) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg E4/3 mg DRSP (N=1864)
Urinary tract infection (Infections and infestations) | 64 (71)
Upper respiratory tract infection (Infections and infestations) | 62 (65)
Viral upper respiratory tract infection (Infections and infestations) | 61 (71)
Bacterial vaginosis (Infections and infestations) | 45 (47)
Sinusitis (Infections and infestations) | 29 (30)
Fungal infection (Infections and infestations) | 24 (32)
Influenza (Infections and infestations) | 24 (27)
Vulvovaginal mycotic infection (Infections and infestations) | 24 (27)
Pharyngitis streptococcal (Infections and infestations) | 18 (20)
Metrorrhagia (Reproductive system and breast disorders) | 86 (88)
Dysmenorrhoea (Reproductive system and breast disorders) | 66 (69)
Breast tenderness (Reproductive system and breast disorders) | 54 (55)
Vaginal haemorrhage (Reproductive system and breast disorders) | 41 (45)
Menorrhagia (Reproductive system and breast disorders) | 39 (40)
Breast pain (Reproductive system and breast disorders) | 26 (27)
Vaginal discharge (Reproductive system and breast disorders) | 20 (20)
Nausea (Gastrointestinal disorders) | 70 (74)
Abdominal pain (Gastrointestinal disorders) | 39 (43)
Vomiting (Gastrointestinal disorders) | 29 (31)
Diarrhoea (Gastrointestinal disorders) | 24 (24)
Abdominal distension (Gastrointestinal disorders) | 20 (20)
Abdominal pain lower (Gastrointestinal disorders) | 18 (18)
Anxiety (Psychiatric disorders) | 45 (45)
Mood swings (Psychiatric disorders) | 38 (40)
Depression (Psychiatric disorders) | 35 (38)
Libido decreased (Psychiatric disorders) | 25 (25)
Insomnia (Psychiatric disorders) | 22 (23)
Mood altered (Psychiatric disorders) | 19 (19)
Irritability (Psychiatric disorders) | 18 (18)
Headache (Nervous system disorders) | 94 (100)
Dizziness (Nervous system disorders) | 22 (23)
Weight increased (Investigations) | 62 (62)
Acne (Skin and subcutaneous tissue disorders) | 63 (69)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (33)
Fatigue (General disorders) | 42 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT02817841/SAP_000.pdf
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02817841/Prot_001.pdf